CLINICAL TRIAL: NCT01589861
Title: A Phase Ib/II Open-label Study Evaluating Safety and Efficacy of Oral BKM120 in Combination With Lapatinib in HER2+/PI3K-activated, Trastuzumab-resistant Locally Advanced, Recurrent and Metastatic Breast Cancer. PIKHER2/IPC 2011-001
Brief Title: Safety and Efficacy of BKM120 and Lapatinib in HER2+/PI3K-activated, Trastuzumab-resistant Advanced Breast Cancer
Acronym: PIKHER2
Status: Suspended | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Data analysis
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PIKHER2/IPC 2011-001
Record Dates: First submitted 2012-03-28; First posted 2012-05-02 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — NVP-BKM120; Lapatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BKM120+Lapatinib (Experimental): BKM120 40, 60 or 80 mg/day per os for 28 days cycle
  + Lapatinib 750, 1000 or 1250 mg/day per os for 28 days cycle
  Interventions: Drug: BKM120 + lapatinib

INTERVENTIONS:
Drug: BKM120 + lapatinib — BKM120 40, 60 or 80 mg/day per os for 28 days cycle associated to lapatinib 750, 1000 or 1250 mg/day per os for 28 days cycle until progression or toxicity
  Other Names: BKM120 and lapatinib

SUMMARY:
This study is based upon the following points:

1. Resistance to trastuzumab, either primary or secondary, is a clinically relevant issue.
2. PI3K/AKT activation, due to loss of expression/function of PTEN and/or activating mutations of PIK3CA, is a mechanism of resistance with clinical relevance in breast cancer. Such activation can be detected by:

   * IHC evaluation of PTEN protein expression
   * genotyping of PIK3CA exon 9 and 20
   * IHC evaluation of phospho-AKT expression
3. BKM120 is an effective PI3K inhibitor. BKM120 and anti-HER2 therapy may have a synergistic antitumor activity in preclinical model of HER2+ breast cancer.
4. Lapatinib is an effective anti-HER2 therapy in trastuzumab-resistant disease.
5. For the evaluation of novel targeted therapies, selecting a patient population enriched for activation of the target to be modulated should allow to maximize the differences in clinical outcome that are expected in the experimental arm, and thus to minimize the patient number to include.
6. We propose to test in a phase I/II study the combination of lapatinib and BKM120 in trastuzumab-resistant HER2+ MBC patients, enriched for activation of PI3K/AKT as detected by loss of expression of PTEN (IHC), and/or mutation of PIK3CA and/or overexpression of phospho-AKT (IHC). Only for phase II patients, mutational status will be an inclusion criteria. For phase I patients molecular status will be a retrospective exploratory analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Female or male ≥ 18 years
2. WHO performance status ≤ 1
3. Locally advanced, recurrent or metastatic, histologically confirmed HER2 positive (IHC 3+ or FISH positive) breast cancer after failure of trastuzumab treatment.

   while on trastuzumab or within 4 weeks since the last infusion of trastuzumab for metastatic disease within 12 months of the last infusion for patients who received trastuzumab as adjuvant or neoadjuvant treatment
4. For the phase II part, progression on trastuzumab must have occurred within 16 weeks before entering this trial.
5. should not have received more than 3 lines of anti-HER2 therapy.
6. For the phase II part, activation of PI3K/AKT pathway
7. capable of understanding the protocol and has signed the informed consent
8. laboratory values within normal range
9. Measurable disease
10. Patients may have received treatment for brain metastases, but must be neurologically stable
11. Baseline LVEF>50% (MUGA or ECHO)
12. Affiliation to social security

Exclusion Criteria:

1. Previous treatment with lapatinib, neratinib or a PI3K inhibitor
2. untreated brain metastases.
3. acute or chronic liver, renal disease or pancreatitis
4. any peripheral neuropathy ≥ CTCAE grade 2
5. any of the following mood disorders, or meets the cut-off score of ≥ 10 in the PHQ-9 or a cut-off of ≥ 15 in the GAD-7 mood scale, respectively, or selects a positive response of '1, 2, or 3' to question number 9 regarding potential for suicidal thoughts ideation in the PHQ-9 (independent of the total score of the PHQ-9)

   * Medically documented history of or active major depressive episode, bipolar disorder (I or II), obsessive-compulsive disorder, schizophrenia, a history of suicidal attempt or ideation, or homicidal ideation (immediate risk of doing harm to others)
   * ≥ CTCAE grade 3 anxiety
6. diarrhea ≥ CTCAE grade 2
7. active cardiac disease
8. history of cardiac dysfunction
9. poorly controlled diabetes mellitus (HbA1c > 8 %)
10. Other severe and/or uncontrolled concomitant medical conditions
11. Impairment of gastrointestinal function that may significantly alter the absorption of BKM120
12. been treated with any hematopoietic colony-stimulating growth factors ≤ 2 weeks prior to starting study drug.
13. currently receiving treatment with medication with a known risk prolong the QT interval or inducing Torsades de Pointes
14. currently being treated with drugs known to be moderate and strong inhibitors or inducers of isoenzyme CYP3A
15. receiving chronic treatment with steroids or another immunosuppressive agent.
16. have received chemotherapy or targeted anticancer therapy ≤ 4 weeks (6 weeks for nitrosourea, antibodies [other than trastuzumab] or mitomycin-C) prior to starting study drug or who have not recovered from side effects of such therapy
17. have received small molecule therapeutics (excluding monoclonal antibodies) ≤ 5 effective half lives prior to starting study drug or who have not recovered from side effects of such therapy
18. have received wide field radiotherapy ≤ 4 weeks or limited field radiation for palliation ≤ 2 weeks prior to starting study drug or who have not recovered from side effects of such therapy
19. have undergone major surgery ≤ 28 days prior to starting study drug or who have not recovered from side effects of such therapy
20. Known diagnosis of HIV infection
21. History of another malignancy within 3 years
22. Patient is unable or unwilling to abide by the study protocol
23. pregnant or breast feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2011-12; Primary Completion 2018-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Phase Ib: maximum-tolerated dose (MTD) | Day 28
  To determine the maximum-tolerated dose (MTD) of BKM120 when administered orally in combination with daily lapatinib to adult patients trastuzumab-resistant HER2+ locally advanced, recurrent and metastatic breast cancer.
Phase II: objective response rate (ORR) | until progression assessed up to 1 year
  To determine the efficacy of daily BKM120 in combination with daily lapatinib as measured by objective response rate (ORR), defined by complete response (CR) or partial response (PR) of target and non target lesions according to RECIST V1.1., in patients with activation of PI3K/AKT pathway detected according to one at least of the following criteria, measured on primary or metastatic tissue: PTEN negative by IHC and/or somatic mutations (exons 9 and 20) of PIK3CA and/or Overexpression of phospho-AKT by IHC.

SECONDARY OUTCOMES:
safety | until progression or end of treatment assessed up to 1 year
  Number of patients with adverse events (according to CTCAE V4)
clinical benefit (CB) | until progression assessed up to 1 year
  - To evaluate clinical benefit (CB defined as complete response (CR) + partial response (PR) + Stable disease (SD) > 6 months)
progression-free survival (PFS) | until progression assessed up to 1 year
  - To assess progression-free survival (PFS)
pharmacokinetics | D1, D8, D15, D22, D28 post dose
  - To determine pharmacokinetics profile (CMax, AUC) of oral BKM120 in combination with orally lapatinib and to monitor exposure to lapatinib

CONTACTS AND LOCATIONS:
Overall Officials: Anthony GONCALVES, MD PhD, Principal Investigator — Institut Paoli-Calmettes
Locations (1):
- Institut Paoli-Calmettes, Marseille, France

REFERENCES:
- [Derived] Guerin M, Rezai K, Isambert N, Campone M, Autret A, Pakradouni J, Provansal M, Camerlo J, Sabatier R, Bertucci F, Charafe-Jauffret E, Hervieu A, Extra JM, Viens P, Lokiec F, Boher JM, Goncalves A. PIKHER2: A phase IB study evaluating buparlisib in combination with lapatinib in trastuzumab-resistant HER2-positive advanced breast cancer. Eur J Cancer. 2017 Nov;86:28-36. doi: 10.1016/j.ejca.2017.08.025. Epub 2017 Sep 23. PMID 28950146
- See also: official web site of the sponsor — http://institutpaolicalmettes.fr